CLINICAL TRIAL: NCT04486378
Title: A Multi-site, Open-label, Phase II, Randomized, Controlled Trial to Compare the Efficacy of RO7198457 Versus Watchful Waiting in Resected, Stage II (High Risk) and Stage III Colorectal Cancer Patients Who Are ctDNA Positive Following Resection
Brief Title: A Phase II Clinical Trial Comparing the Efficacy of RO7198457 Versus Watchful Waiting in Patients With ctDNA-positive, Resected Stage II (High Risk) and Stage III Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT122-01; 2020-000451-12 (EudraCT Number); U1111-1250-5294 (Other: WHO Universal Trial Number (UTN)); 2023-509516-28-00 (EU CTIS Number)
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer Stage II; Colorectal Cancer Stage III
Keywords: Cancer; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- RO7198457 (Experimental): Participants will receive a recommended dose of RO7198457.
  Interventions: Drug: RO7198457 intravenous (IV)
- Observational Group (Other): Observational group will undergo watchful waiting, which is the standard of care in this setting.
  Interventions: Other: Observational group (no intervention)
- Biomarker Cohort (Experimental)
  Interventions: Drug: RO7198457 intravenous (IV)
- Exploratory Cohort (Experimental)
  Interventions: Drug: RO7198457 intravenous (IV)
- Colorectal Liver Metastasis (CLM) Cohort (Experimental)
  Interventions: Drug: RO7198457 intravenous (IV)

INTERVENTIONS:
Drug: RO7198457 intravenous (IV) — RO7198457 administered as an IV injection at protocol-specified intervals over 12 months.
  Arms: Biomarker Cohort; Colorectal Liver Metastasis (CLM) Cohort; Exploratory Cohort; RO7198457
Other: Observational group (no intervention) — watchful waiting
  Arms: Observational Group

SUMMARY:
This is a multi-site, open-label, Phase II, randomized, trial to compare the efficacy of RO7198457 versus watchful waiting in patients with circulating tumor DNA (ctDNA) positive, surgically resected Stage II/III rectal cancer, or Stage II (high risk)/Stage III colon cancer.

DETAILED DESCRIPTION:
Patients will receive up to 15 doses of RO7198457 over the course of trial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be a man or woman of at least 18 years of age.
* Patients must have Stage II/Stage III rectal cancer or Stage II (high risk)/Stage III colon cancer per American Joint Committee on Cancer (AJCC) 2017 that has been surgically totally resected (R0 confirmed by pathology report). Stage II (high risk) colon cancer is defined as Stage II disease with any of the following risk factors for recurrence:

  * T4
  * Grade ≥ 3.
  * Clinical presentation with bowel obstruction or perforation.
  * Histological signs of vascular, lymphatic or perineural invasion.
  * < 12 nodes evaluated after surgery.

    * For the CLM Cohort: patients must have metastatic colorectal cancer (mCRC) (Stage IV) with resected CLM (synchronous and metachronous CLM within 6 months of initial diagnosis) per AJCC 2017, after standard of care (SoC) primary resection and curative-intent hepatectomy (R0 confirmed by pathology report) with or without (neo-)adjuvant chemotherapy (prior to hepatectomy), and planned adjuvant chemotherapy.
    * For the Biomarker Cohort: patients with tumors of the colon, including but not limited to, colon adenocarcinoma, carcinoid tumors (including goblet cell carcinoid/adenocarcinoma), and tumors of the appendix, whose tumors were surgically resected and are planned for adjuvant chemotherapy (per institutional standards), can be included.
* Patients must have detectable ctDNA prior to start of adjuvant chemotherapy (AdCTx) (except for the Biomarker Cohort).

  * ctDNA assay must be performed through this trial or study BNT000-001 ctDNA screening protocol.
* Patients must have an Eastern Cooperative Oncology Group Performance Status of 0-1.
* Patients must have adequate hematologic, bone marrow and organ function as defined by the protocol.
* Adequate tumor material in formalin-fixed paraffin embedded blocks or as sectioned tissue (only upon approval by sponsor) must be available (as described in the laboratory manual). For the CLM Cohort: tumor material must come from primary resection for patients who undergo staged approach, or from available archival material from the previously untreated tumor biopsy from the primary.
* At least 5 tumor neoantigens identified in the provided tumor sample.
* The patient has started a standard of care AdCTx preferably within 8 weeks but no later than 10 weeks post-surgery and has completed at least 3 months of treatment of a 3- or a 6-month course of chemotherapy (including rest days). For the CLM Cohort: patient must have completed AdCTx with or without (neo-)adjuvant chemotherapy for up to 6 months in total or total intended amount determined by care providers per SoC. AdCTx must have started preferably within 8 weeks, but no later than 10 weeks, after hepatectomy. For the Biomarker Cohort: patient must have received at least one cycle of adjuvant chemotherapy per institutional standards.

Exclusion Criteria:

* Patients with uncontrolled intercurrent illness as defined by the protocol.
* Diagnosed microsatellite instability high tumors.
* Prior therapy with any of the following:

  * Neo-adjuvant (radio)chemotherapy prior to surgery.
  * Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of trial treatment or anticipation of need for systemic immunosuppressive medication during trial treatment, with the exception of low dose steroids defined as 10 mg oral prednisone (or equivalent).
  * Current or recent (within the 28 days prior to randomization) treatment with another investigational drug.

    * Exception for the CLM Cohort: primary tumor must be resected and (neo-)adjuvant chemotherapy prior to curative-intent hepatectomy is accepted.
* Toxicities from previous anti-cancer therapies that have not resolved to baseline levels or to Grade 1 or less except for alopecia and peripheral neuropathy.
* Patients who developed metastatic disease during screening/receiving standard of care treatment (not applicable for the Exploratory Cohort or the Biomarker Cohort).
* Patients with known past or current malignancy other than inclusion diagnosis, except for:

  * Cervical carcinoma of Stage 1B or less.
  * Non-invasive basal cell or squamous cell skin carcinoma.
  * Non-invasive, superficial bladder cancer.
  * Prostate cancer with a current prostate-specific antigen level < 0.1 ng/mL.
  * Any curable cancer with a complete response of > 2 years duration.
* Patients with known allergies, hypersensitivity, or intolerance to RO7198457 or its excipients.
* Patients who had major surgery (e.g., surgery requiring general anesthesia) within 4 weeks before screening, or will not have fully recovered from surgery, or have surgery planned during the time the patient are expected to participate in the trial.
* Patients with positive serology for hepatitis B indicative of active hepatitis B infection:

  * Positive test for hepatitis B surface antigen (HBsAg) OR
  * Negative test for HBsAg AND positive test for antibodies to hepatitis B core antigens (anti-HBc) AND positive test for hepatitis B virus (HBV) DNA.

    * Serological markers indicative of vaccination (isolated antibodies to hepatitis B surface antigens [anti-HBs]) or resolved natural infection without viral load (anti-HBc with negative HBsAg and negative HBV DNA) are not exclusionary.
* Active Hepatitis C virus (HCV) infection; patients who have completed curative antiviral treatment with HCV viral load below the limit of quantification are allowed.
* Patients who have a history of human immunodeficiency virus (HIV) antibody positivity, or tests positive for HIV at screening.
* Patients who have had prior splenectomy.

NOTE: Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Through study completion, up to 5 years
  DFS defined as the time from randomization to occurrence of any of the following events, whichever occurs first:
  * Locoregional recurrence or distant metastases as determined by an independent central radiology assessment.
  * Occurrence of second primary (same or other) cancer as determined by an independent central radiology assessment.
  * Death from any cause.
  * Loss to follow-up is censored.

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | Through study completion, up to 5 years
  RFS is defined as the time from randomization to occurrence of any of the following events, whichever occurs first:
  * Locoregional recurrence or distant metastases as determined by the investigator.
  * Death from any cause.
  * Occurrence of second primary (same or other) cancer as determined by the investigator is ignored.
  * Loss to follow-up is censored.
Time to recurrence (TTR) | Through study completion, up to 5 years
  TTR is defined as the time from randomization to occurrence of any of the following events (i.e., events related to the same cancer), whichever occurs first:
  * Locoregional recurrence or distant metastases as determined by the investigator.
  * Death from same cancer.
  * Occurrence of second primary (same or other) cancer as determined by the investigator is ignored.
  * Loss to follow-up and deaths from other cancer, non-cancer-related deaths, treatment-related deaths are censored.
Time to treatment failure (TTF) | Through study completion, up to 5 years
  TTF is defined as the time from randomization to occurrence of any of the following events, whichever occurs first:
  * Locoregional recurrence or distant metastases as determined by the investigator.
  * Occurrence of second primary (same or other) cancer as determined by the investigator.
  * Death from any cause except non-cancer related death.
  * Start of new cancer therapy.
  * Loss to follow-up and non-cancer-related deaths are censored.
Overall survival (OS) | Through study completion, up to 5 years
  OS defined as the time from randomization to death from any cause.
Change of ctDNA status (approximately every 3 months) | Through study completion, up to 5 years
Occurrence of treatment emergent adverse event (TEAE) | 15 months
  TEAE, including Grade 3+, serious, fatal TEAE by relationship (adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0).
Occurrence of dose reduction and discontinuation of RO7198457 due to a TEAE. | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (121):
- United States (39):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - John Muir Clinical Research Center, Concord, California
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - Marin Cancer Care, Greenbrae, California
  - St Joseph Hospital of Orange, Orange, California
  - Sansum Clinic, Santa Barbara, California
  - Rocky Mountain Cancer Centers - Denver Midtwon, Denver, Colorado
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Florida Cancer Specialist South, Fort Myers, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Cancer Care Center of Decatur, Cancer Care Specialists of IL, Decatur, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - Josephine Ford Cancer Center-Henry Ford Cancer Center, Detroit, Michigan
  - Allina Health, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - New York Oncology Hematology, P.C., Albany, New York
  - Weill Cornell Medical College, New York, New York
  - New York - Presbyterian Hospital - Columbia University Medical center, New York, New York
  - Oncology Hematology Care Clinical Trials, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center Medical University Of South Carolina, Charleston, South Carolina
  - Sarah Cannon (Tennessee Oncology - Nashville), Nashville, Tennessee
  - Sarah Cannon Research Institute (SCRI) Oncology Partners, Nashville, Tennessee
  - Texas Oncology, P.A. - Austin, Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology-San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - University of Washington, Seattle, Washington
  - MultiCare Institute for Research & Innovation, Spokane, Washington
  - Northwest Cancer Specialists P.C., Vancouver, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (10):
  - Imeldaziekenhuis General Hospital, Bonheiden
  - VZW Algemeen Ziekenhuis AZ Klina, Brasschaat
  - Institut Jules Bordet, Brussels
  - GHDC (Grand Hopital de Charleroi), Charleroi
  - AZ Groeninge, Kortrijk
  - Centres Hospitaliers Jolimont, La Louvière
  - Universitaire Ziekenhuizen Leuven, Leuven
  - AZ Delta Roeselare, Roeselare
  - GasthuisZusters Antwerpen - Sint-Augustinus, Wilrijk
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa
  - Princess Margaret Cancer Centre, Toronto
- Germany (24):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitaetsklinikum St. Josef-Hospital Bochum, Bochum
  - Universitätsklinikum Bonn, Med. Klinik u. Poliklinik I, Bonn
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Krankenhaus Nordwest GmbH - Institut Fuer Klinisch-Onkologische Forschung (IKF), Frankfurt am Main
  - Klinikum der Johann Wolfgang Goethe-Universitaet Frankfurt, Frankfurt am Main
  - Studiengesellschaft BSF, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Hämatologisch-Onkologische Praxis Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - National Center for Tumor Diseases (NCT) Heidelberg, Heidelberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Staedtisches Krankenhaus Kiel gGmbH, Kiel
  - Universitaetsklinikum Leipzig AoeR, Leipzig
  - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz KoeR, Mainz
  - Klinikum der Philipps-Universität Marburg, Marburg
  - LMU Klinikum (Campus Großhadern) Medizinische Klinik Universität München, München
  - Städtisches Klinikum München GmbH, Klinikum Neuperlach, München
  - OhO Ostholstein Onkologie, Oldenburg in Holstein
  - Prosper Hospital, Recklinghausen
  - Robert-Bosch-Krankenhaus - Centrum fuer Tumorerkrankungen, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Spain (25):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Nuestra Senora de Sonsoles, Ávila
  - Hospital Universitari Germans Trias - ICO Badalona, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Clinic Hematolo/Oncologia- ICMHO, Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Clinica Universidad Navarra, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HMN Sanchinarro, Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Hospital Regional Universitario Carlos Haya Malaga - Instituto de Investigacion Biomedica de Malaga, Málaga
  - Complejo Hospitalario de Orense, Ourense
  - Clinica Universitaria de Navarra, Pamplona
  - Complejo Hospitalario de Navarra (CHN), Pamplona
  - Hospital Universitario Marques De Valdecilla, Santander
  - Complejo Hospitalario Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio - Hospital de la Mujer, Seville
  - Consorcio Hospital General Valencia, Valencia
  - Complexo Hospitalario Universitario de Vigo (CHUVI), Vigo
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (3):
  - Lunds Universitet - Medicinska Fakulteten (Lund University Faculty of Medicine), Lund
  - Sodersjukhuset, Onkologiska Kliniken, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
- United Kingdom (18):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington
  - Queen Elizabeth Hospital Birmingham-University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Velindre NHS Trust, Velindre Cancer Centre, Cardiff
  - Hull and East Yorkshire Hospitals NHS Trust - Castle Hill Hospital, Cottingham
  - Dorset County Hospital NHS Foundation Trust - Dorset County Hospital, Dorchester
  - Beatson West of Scotland Cancer Centre - Gartnavel Royal Hospital - NHS Greater Glasgow and Clyde, Glasgow
  - St Bartholomew's Hospital-Barts Health NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Guy's and St Thomas' Hospital NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust- Chelsea, London
  - The Christie NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne
  - Churchill Hospital - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Royal Preston Hospital - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - University Hospital Southampton NHS Foundation Trust - Southampton General Hospital, Southampton
  - The Royal Marsden NHS Foundation Trust, Sutton
  - Torbay Hospital - South Devon Healthcare Nhs Foundation Trust, Lowes Bridge, Torquay

IPD SHARING:
Plan to Share IPD: No